CLINICAL TRIAL: NCT02457910
Title: A Phase Ib/II Trial of Taselisib (GDC-0032), a PI3K Inhibitor, in Combination With Enzalutamide in Patients With Androgen Receptor Positive Triple Negative Metastatic Breast Cancer
Brief Title: Taselisib and Enzalutamide in Treating Patients With Androgen Receptor Positive Triple-Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim analysis - toxicity
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Translational Breast Cancer Research Consortium (Other); Conquer Cancer Foundation (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Vandana Abramson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 1374; NCI-2015-00795 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GO28972; TBCRC 032; VICC BRE 1374 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-29 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; Progesterone Receptor Negative; Progesterone Receptor Positive; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — enzalutamide; 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Taselisib 2 mg (Experimental): Patients receive taselisib PO QD on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study; Drug: Taselisib
- Enzalutamide (Active Comparator): Patients receive enzalutamide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients may crossover to receive Enzalutamide + Taselisib
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study
- Taselisib 4 mg (Experimental): Patients receive taselisib PO QD on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study; Drug: Taselisib
- Taselisib 6 mg (Experimental): Patients receive taselisib PO QD on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study; Drug: Taselisib
- Taselisib 8 mg (Experimental): Patients receive taselisib PO QD on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study; Drug: Taselisib
- Enzalutamide + Taselisib (Experimental): Patients receive enzalutamide PO QD starting on day 1 of cycle 1, and will receive Taselisib PO QD starting on day 1 of cycle 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study; Drug: Taselisib
- Cross-Over (Experimental): Upon progression of disease, patients on the enzalutamide only arm will be allowed to crossover to enzalutamide + taselisib (must begin no later than 21 days after the clinic visit at which disease progression is determined) Enzalutamide and Taselisib will be taken PO QD
  Interventions: Other: Biomarker Analysis; Drug: Enzalutamide; Other: Pharmacological Study; Drug: Taselisib

INTERVENTIONS:
Other: Biomarker Analysis — Correlative studies
Drug: Enzalutamide — Given PO
  Other Names: MDV3100; Xtandi
Other: Pharmacological Study — Correlative studies
Drug: Taselisib — Given PO
  Other Names: GDC-0032
  Arms: Cross-Over; Enzalutamide + Taselisib; Taselisib 2 mg; Taselisib 4 mg; Taselisib 6 mg; Taselisib 8 mg

SUMMARY:
This partially randomized phase Ib/II trial studies the side effects and best dose of taselisib when given together with enzalutamide and to see how well they work in treating patients with androgen receptor positive triple-negative breast cancer that has spread to other places in the body. Taselisib is a PI3K inhibitor. The PI3K pathway is involved is cancer growth. Androgen may cause the growth of tumor cells. Enzalutamide may stop the growth of tumor cells by blocking the androgen receptor from working. Giving taselisib with enzalutamide may be a better treatment for patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of taselisib given in combination with enzalutamide: Assessment of dose limiting toxicities (DLTs) during the first 4 weeks of treatment (cycle 1). (Phase Ib) II. To determine the safety and tolerability of taselisib given in combination with enzalutamide: Determination of the maximally tolerated dose (MTD) of taselisib given in combination with enzalutamide. (Phase Ib) III. To evaluate the efficacy, as measured by clinical benefit rate (CBR), of enzalutamide + taselisib in patients with androgen receptor positive (AR+) triple negative (TN) metastatic breast cancer (MBC). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the progression free survival (PFS) of enzalutamide + taselisib in patients with AR+ TN MBC.

II. To assess the pharmacokinetics (PKs) of taselisib and enzalutamide in patients with AR+ TN MBC.

TERTIARY OBJECTIVES:

I. To explore predictors of biomarker response and mechanisms of resistance based on exploratory analysis of tumor tissue obtained through biopsies.

II. Levels of phosphatase and tensin homolog (PTEN) expression by immunohistochemistry (IHC) and quantitative real-time polymerase chain reaction (qPCR).

III. Presence of mutations in the phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) gene.

IV. Human epidermal growth factor receptor 2 (HER2) (IHC, fluorescence in situ hybridization [FISH]) and estrogen receptor (ER)/progesterone receptor (PR) levels (IHC) in tumor biopsy from a metastatic site.

V. Levels of mitogen-activated protein kinase kinase (MEK) activity measured by phosphorylated extracellular-signal-regulated kinases (p-ERK1/2) (IHC) and phosphorylated p-ribosomal protein S6 (S6) (S235/236 and S240/244) at baseline and upon progression of disease.

VI. Levels of phosphorylated v-akt murine thymoma viral oncogene homolog 1 (p-AKT) (IHC) at baseline and upon progression of disease.

VII. Gene expression profiling to assign a triple negative subtype. VIII. Whole exome deoxyribonucleic acid (DNA)-sequencing (seq) on DNA isolated at baseline and upon progression.

IX. Plasma for circulating tumor DNA (ctDNA) analysis to assess PIK3CA mutation status in response and resistance.

X. To assess the predictive effects of PIK3CA mutations and PTEN loss on PFS and CBR.

XI. To evaluate the ability of multi-parametric magnetic resonance imaging (MRI) performed early in therapy to predict both biological and clinical response.

OUTLINE: This is a phase Ib, dose-escalation study of taselisib followed by a randomized phase II study.

PHASE IB: Patients receive taselisib orally (PO) once daily (QD) on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive taselisib PO QD and enzalutamide as in Phase Ib. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.

ARM II: Patients receive enzalutamide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients may crossover to Arm I.

After completion of study treatment, patients are followed up for 30 days and then every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide informed written consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Clinical stage IV invasive mammary carcinoma
* For phase 1b: HER2 negative, as defined for phase II; any ER/PR (negative or positive) can be enrolled in the phase 1b portion
* For phase II: ER negative (defined as expression of ER in =< 1% cells), PR negative (defined as expression of PR in =< 1% cells), HER2 negative (acceptable methods of HER2 analysis include IHC [0, 1+], fluorescence in situ hybridization [FISH] with HER2/centromere on chromosome 17 [CEN17] ratio < 2, and/or chromogenic in situ hybridization [CISH] with HER2/CEN-17 ratio < 2), as previously documented by histological analysis
* Androgen receptor positivity, defined as >= 10% of tumor cell nuclei with immunoreactivity for AR on central review at Vanderbilt
* Measurable or bone-only evaluable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension by Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1, with radiologic scans within 21 days of day 1, cycle 1
* Any number of prior therapies as long as patients have adequate performance status and meet all other eligibility criteria
* Prior treatment with anti-androgens other than enzalutamide is acceptable
* Phase 1b only: Formalin-fixed paraffin embedded blocks (FFPB) or fresh frozen tissue from the original diagnosis or the metastatic setting should be located; tissue must be submitted with 3 weeks of study initiation
* Phase II only: Biopsy of a metastatic lesion in patients with reasonably accessible metastatic lesions (chest wall, skin, subcutaneous tissue, lymph nodes, skin, breast, bones, lung, and liver metastases); if a reasonably accessible metastatic lesion is not available, the patient may go on study provided that archived tissue is available; however, if a reasonably accessible site is available for biopsy, the patient must agree to biopsy; any patients not undergoing biopsy must be approved for study enrollment by the Protocol Chair; biopsies may be done with local anesthesia or intravenous conscious sedation, according to institutional guidelines; if a biopsy requires general anesthesia, then it is only allowed if acquisition of tissue is clinically indicated, and excess tissue may be collected for research purposes; patients without sites available for biopsy must have available tissue (archived formalin-fixed paraffin embedded blocks [FFPB] or fresh frozen tissue from original diagnosis or metastatic setting) for correlative studies; tissue needs to be located and available at the time of registration (tissue needs to be submitted within 3 weeks of study initiation)
* Patients must have adequate hematologic, hepatic, and renal function. All tests must be obtained within 28 days of starting treatment. Labs are to be repeated on cycle 1, day 1 and must still meet eligibility. These include:
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin (HgB) >= 9 g/dL
* Creatinine =< 1.5 X upper limits of normal (ULN)
* international normalized ratio (INR) ≤2
* Total serum bilirubin =< 1.5 x ULN (in patients with known Gilbert syndrome, a total bilirubin =< 3.0 x ULN, with direct bilirubin =< 1.5 x ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (or =< 5.0 x ULN if hepatic metastases are present)
* For patients without known type II diabetes, the following is required at screening:

  * Fasting plasma glucose =< 160 mg/dL (7.49 mmol/L) and glycosylated hemoglobin (HbA1c) < 7.5 % or International Federation of Clinical Chemistry (IFCC) < 53 mmol/mol
* For patients with type II diabetes receiving only oral anti-hyperglycemic therapy (patients receiving insulin are not eligible), the following are required at screening:

  * HbA1c < 8.5 % or IFCC < 69.4 mmol/mol
  * Stable regimen of oral anti-hyperglycemic therapy without insulin usage for at least 3 weeks prior to first study treatment
  * Fasting plasma glucose levels =< 160 mg/dL (8.88 mmol/L) and no hypoglycemia (blood sugar [BS] < 60) during home monitoring for at least 1 week prior to study entry
* Patients must be able to swallow and retain oral medication
* For patients who are not postmenopausal or surgically sterile (absence of ovaries and/or uterus), agreement to remain abstinent or to use two adequate methods of contraception (e.g., condoms, diaphragm, vasectomy/vasectomized partner, tubal ligation), during the treatment period and for at least 30 days after the last dose of study treatment or 3 months after discontinuation of taselisib and/or enzalutamide, whichever is longer; hormone based oral contraceptives are not allowed on study; postmenopausal is defined as:

  * Age >= 60 years
  * Age =< 60 years and amenorrheic for 12 months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression; or follicle stimulating hormone and estradiol in the postmenopausal range
* Patients may have received radiation therapy to painful bone metastases or areas of impending bone fracture as long as radiation therapy is completed >= 2 weeks prior to day 1 of cycle 1 of treatment; patients who have received prior radiotherapy must have recovered from toxicity (=< grade 1) induced by this treatment; baseline radiologic scans must be obtained after completion of radiation
* Patients must complete all screening assessments

Exclusion Criteria:

* Any kind of malabsorption syndrome significantly affecting gastrointestinal function, including history of Crohn's disease or inflammatory bowel disease
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, biologic therapy) other than the ones specified in the protocol; patients must have discontinued the above cancer therapies for 1 week prior to the first dose of study medication, as well as recovered to baseline from toxicity induced by previous treatments; any investigational drugs should be discontinued 2 weeks prior to the first dose of study medication and radiotherapy must have been completed >= 2 weeks prior to initiation of study drug (cycle 1, day 1)
* Prior use of PI3K or Akt inhibitors in the metastatic setting for the treatment of cancer; these include, but are not limited to: taselisib, GDC-0941, GDC-0980, BEZ235, BKM120, LY294002, PIK-75, TGX-221, XL147, XL765, SF1126, PX-866, D-87503, D-106669, GSK615, CAL101; patients who have received PI3K/Akt inhibitors previously for < 4 weeks will be eligible
* Prior treatment with enzalutamide
* Current or previously treated brain metastasis or active leptomeningeal disease; head imaging is required during screening in all patients to exclude the presence of central nervous system (CNS) metastatic disease
* History of seizure or any condition that may predispose to seizure; history of loss of consciousness or transient ischemic attack within 12 months before day 1
* Pregnant or lactating women
* Insulin-dependent diabetes; patients with type II diabetes must meet the inclusion criteria outlined above
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring parenteral antibiotics
  * Impairment of lung function (chronic obstructive pulmonary disease [COPD] > grade 2, lung conditions requiring oxygen therapy) or current dyspnea at rest
  * Symptomatic congestive heart failure (class III or IV of the New York Heart Association classification for heart disease)
  * Known left ventricular ejection fraction (LVEF) < 50%
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * Uncontrolled hypertension (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg, found on two consecutive measurements separated by a 1 or 2-week period despite adequate medical support)
  * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [National Cancer Institute-Common Terminology Criteria for Adverse Events, version 4.0, grade 3])
  * Corrected QT using the Fridericia correction formula (QTcF) >= 480 msec on screening electrocardiogram (EKG)
  * Known history of QT/correct QT (QTc) prolongation or Torsades de Pointes (TdP)
  * ST depression or elevation of >= 1.5 mm in 2 or more leads
  * Diarrhea of any cause >= Common Terminology Criteria for Adverse Events (CTCAE) grade 2
  * Active autoimmune disease that is not controlled by nonsteroidal or steroidal (< 10 mg of prednisone per day) anti-inflammatory drugs or active inflammatory disease, including small or large intestine inflammation such as active Crohn's disease or ulcerative colitis, which requires immunosuppressive therapy
  * Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary
  * Known history of chronic liver disease including cirrhosis, current alcohol abuse, or infection with hepatitis B virus or hepatitis C virus (active or carrier) or renal failure
  * Known history of chronic pancreatitis
  * Conditions that affect lymphocyte counts, such as human immunodeficiency virus (HIV) infection or immunosuppressive therapy
* Use of prohibited drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Abramson, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (12):
- United States (12):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - John Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor Breast Center, Houston, Texas

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 enrolled in Phase Ib and 17 in phase II
Pre-assignment Details: 13 in phase Ib and 17 in phase II
Groups:
- PH1b E+T - Level 1 (Cohort 1): Enzalutamide 160 mg PO daily and 2 mg Taselisib PO daily
- PH1b E+T - Level 2 (Cohort 1 and 2): Enzalutamide 160 mg PO daily and Taselisib 4 mg PO daily
- PH1b E+T - Level 3 (Cohort 1): Enzalutamide 160 mg PO daily and Taselisib 6 mg PO daily
- PH1b E+T - Level 4 (Cohort 1): Enzalutamide 160 mg PO daily and Taselisib 8 mg PO daily
- PHII Enzalutamide: Enzalutamide 160mg PO daily
- Phase II E+T: Enzalutamide 160mg PO daily and Taselisib 4 mg PO daily
Period: Overall Study
Arm/Group | PH1b E+T - Level 1 (Cohort 1) | PH1b E+T - Level 2 (Cohort 1 and 2) | PH1b E+T - Level 3 (Cohort 1) | PH1b E+T - Level 4 (Cohort 1) | PHII Enzalutamide | Phase II E+T
Started | 3 | 5 (In dose escalation, two patients receiving the 4 mg dose of taselisib were removed for toxicities) | 3 | 2 | 5 (3 participants crossed over to enzalutamide and taselisib) | 12
Completed | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 3 | 5 | 3 | 2 | 5 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 1 | 1 | 3
Not completed — Disease progression | 3 | 3 | 1 | 1 | 4 | 6
Not completed — Other complicating illness | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ER/PR+ or TNBC AR+ women with breast cancer
Groups:
- PH1b E+T - Level 1 (Cohort 1); PH1b E+T - Level 2 (Cohort 1 and 2); PH1b E+T - Level 3 (Cohort 1); PH1b E+T - Level 4 (Cohort 1); Phase II E+T: Enzalutamide and Taselisib taken daily by mouth
- PHII Enzalutamide: Enzalutamide taken daily by mouth
- Total: Total of all reporting groups
Arm/Group | PH1b E+T - Level 1 (Cohort 1) | PH1b E+T - Level 2 (Cohort 1 and 2) | PH1b E+T - Level 3 (Cohort 1) | PH1b E+T - Level 4 (Cohort 1) | PHII Enzalutamide | Phase II E+T | Total
Number analyzed (Participants) | 3 | 5 | 3 | 2 | 5 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 3 | 2 | 2 | 9 | 22
  >=65 years | 1 | 1 | 0 | 0 | 3 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 2 | 5 | 12 | 29
  Male | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 5 | 3 | 2 | 5 | 11 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) - Phase II
Description: CBR is defined as the proportion of patients with a best response of complete response (CR), partial response (PR), or (SD) stable disease per RECIST criteria 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. It is calculated as the mean of binomial distribution.
Time Frame: At 16 weeks
Population: Evaluable TNBC patients who had at least one cycle of treatment and had their disease re-evaluated at 16 weeks or progressed prior to the 16-week assessment
Measure: Mean (95% Confidence Interval); unit: proportion of patients
Groups:
- Arm I (Taselisib, Enzalutamide): Patients receive taselisib PO QD on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
- Arm II (Enzalutamide): Patients receive enzalutamide PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients may crossover to Arm I.
Arm/Group | Arm I (Taselisib, Enzalutamide) | Arm II (Enzalutamide)
Number analyzed (Participants) | 14 | 5
proportion of patients | 0.357 [0.163 to 0.612] | 0 [0 to 0.434]

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Taselisib Combined With 160mg Enzalutamide - Phase I
Description: defined as the highest dose tested in which a dose limiting toxicity is experienced by 0 out of 3 or 1 out of 6 patients among the dose levels. Dose limiting toxicity will be graded according to the National Cancer Institute CTCAE version 4.0.
Time Frame: 4 weeks
Population: 13 patients (7 ER+ and 6 TNBC) breast cancer patients
Measure: Number; unit: DLTs
Groups:
- 2mg Taselisib and 160mg Enzalutamide: Patients receive 2mg taselisib PO QD on days 1-28 and 160mg enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
  160 mg enzalutamide were administered in combination with taselisib starting dose of 2 mg and escalated to 4 mg, 6 mg and 8 mg in a traditional 3+3 trial design.
- 4mg Taselisib and 160mg Enzalutamide: Patients receive 4mg taselisib PO QD on days 1-28 and 160mg enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
- 6mg Taselisib and 160mg Enzalutamide: Patients receive 6mg taselisib PO QD on days 1-28 and 160mg enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
- 8mg Taselisib and 160mg Enzalutamide: Patients receive8mg taselisib PO QD on days 1-28 and 160mg enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
Arm/Group | 2mg Taselisib and 160mg Enzalutamide | 4mg Taselisib and 160mg Enzalutamide | 6mg Taselisib and 160mg Enzalutamide | 8mg Taselisib and 160mg Enzalutamide
Number analyzed (Participants) | 3 | 5 | 3 | 3
DLTs | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Progression-Free Survival (PFS) of Patients Treated With Enzalutamide and Taselisib
Description: The PFS time is defined as the time from treatment start to progression or death (whichever comes first), and those alive without progression were censored at the last date of follow up. PFS will be estimated using the Kaplan-Meier method. The median with 95% confidence intervals will be reported.
Time Frame: Time from course 1, day 1 until objective tumor progression, assessed up to 3 years
Population: Evaluable Androgen Receptor Positive Triple Negative Metastatic Breast Cancer patients that received enzalutamide + taselisib regardless of dose assignment. It is pre-specified by the study protocol to combined groups of TN MBC patients who received both drugs for overall PFS.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Patients Received Both Enzalutamide and Taselisib: Patients received enzalutamide and taselisib from phase I and phase II and evaluable
Arm/Group | Patients Received Both Enzalutamide and Taselisib
Number analyzed (Participants) | 14
months | 3.4 [2.1 to 7.2]

4. Secondary Outcome: Pharmacokinetic Profile
Description: Pharmacokinetic sampling will occur in the phase Ib portion and in 10 patients in the phase II portion
Time Frame: Approximately 4 months
Population: Data was not collected because taselisib is no longer being developed commercially.
Groups:
- Combination of Taselisib and Enzalutamide: Patients receive taselisib PO QD on days 1-28 and enzalutamide PO QD on days 9-28 of course 1 and days 1-28 of subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients experiencing unacceptable toxicity due to enzalutamide may continue to receive taselisib.
  160 mg enzalutamide were administered in combination with taselisib starting dose of 2 mg and escalated to 4 mg, 6 mg and 8 mg in a traditional 3+3 trial design.
Arm/Group | Combination of Taselisib and Enzalutamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 42 months
Groups:
- Enzalutamide + Taselisib: Patients receive enzalutamide PO QD starting on day 1 of cycle 1, and will receive PO QD Taselisib on day 1 of cycle 2.
Arm/Group | Taselisib 2 mg | Taselisib 4 mg | Taselisib 6 mg | Taselisib 8 mg | Enzalutamide | Enzalutamide + Taselisib | Cross-Over
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/5 | 3/3 | 2/2 | 2/2 | 5/12 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/5 | 1/3 | 0/2 | 1/2 | 10/12 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 3/3 | 2/2 | 2/2 | 12/12 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taselisib 2 mg (N=3) | Taselisib 4 mg (N=5) | Taselisib 6 mg (N=3) | Taselisib 8 mg (N=2) | Enzalutamide (N=2) | Enzalutamide + Taselisib (N=12) | Cross-Over (N=3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taselisib 2 mg (N=3) | Taselisib 4 mg (N=5) | Taselisib 6 mg (N=3) | Taselisib 8 mg (N=2) | Enzalutamide (N=2) | Enzalutamide + Taselisib (N=12) | Cross-Over (N=3)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (4) | 2 (4) | 1 (1) | 2 (2) | 7 (7) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (9) | 1 (3) | 2 (4) | 0 (0) | 4 (4) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (15) | 3 (3) | 2 (2) | 0 (0) | 3 (5) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 4 (4) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (4) | 5 (12) | 3 (6) | 2 (2) | 2 (7) | 10 (21) | 3 (3)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 6 (10) | 1 (1)
Limb edema (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (2) | 2 (4) | 0 (0) | 4 (5) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 2 (3)
Alanine amininotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (2)
Weight loss (Investigations) | 2 (2) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (5) | 2 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 0 (0) | 4 (6) | 2 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 0 | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT02457910/Prot_SAP_000.pdf